CLINICAL TRIAL: NCT02717507
Title: Pharmacologic Reversal of Ventricular Remodeling in Childhood Cancer Survivors at Risk for Heart Failure (PREVENT-HF): A Phase 2b Randomized Placebo-Controlled (Carvedilol) Trial
Brief Title: Carvedilol in Preventing Heart Failure in Childhood Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALTE1621; NCI-2016-00232 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE1621 (Other: Children's Oncology Group); COG-ALTE1621 (Other: DCP); ALTE1621 (Other: CTEP); R01CA196854 (NIH); UG1CA189955 (NIH); NCT01347970 (obsolete NCT alias)
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Results first posted 2023-09-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Carvedilol; Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (carvedilol) (Experimental): Patients receive low-dose carvedilol PO QD or BID for 24 months.
  Interventions: Drug: Carvedilol; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD or BID for 24 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Pharmacological Study; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carvedilol — Given PO
  Other Names: Coreg
  Arms: Arm I (carvedilol)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Pharmacological Study — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IIb trial studies how well low-dose carvedilol works in preventing heart failure in cancer survivors exposed to high dose anthracyclines for management of childhood cancer. Patients who received high-dose anthracycline chemotherapy are at a much greater risk for developing heart failure compared to survivors who didn't get any anthracycline chemotherapy. Heart failure happens when the heart muscle has been weakened and can't pump blood as well as it should. Carvedilol may help lower the risk of cardiovascular complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the impact of a two-year course of low-dose carvedilol on surrogate echocardiographic indices of heart failure (HF) risk, including: Left ventricular (LV) posterior wall thickness-dimension ratio (LV T-D); LV systolic and diastolic function, and afterload; Natriuretic peptides, troponins, and galectin-3.

SECONDARY OBJECTIVES:

I. To establish safety and tolerability of this two-year course of low-dose carvedilol, assessing both objective measures (hepatic function) and patient reported outcomes.

II. To examine the modifying effect of demographic, clinical, and molecular characteristics on the risk: benefit ratio from this two-year carvedilol intervention.

EXPLORATORY OBJECTIVE:

I. To evaluate the long-term efficacy of carvedilol in preventing cardiomyopathy and/or heart failure in high-risk childhood cancer survivors.

OUTLINE: This is a dose-escalation study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive low-dose carvedilol orally (PO) once daily (QD) or twice daily (BID) for 24 months.

ARM II: Patients receive placebo PO QD or BID for 24 months.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Males and females must weigh >= 40 Kg
* Patient must have had a cancer diagnosis < 22 years of age, irrespective of current age
* Patient must have a lifetime cumulative anthracycline dose of >= 250 mg/m^2 DOXOrubicin equivalent without the protection of dexrazoxane (Zinecard) therapy; the anthracycline dose threshold must be met as part of the treatment of a cancer that was diagnosed at < 22 years of age

  * Note: Institutional records (e.g., clinic note, treatment summary, chemotherapy roadmap) can be used to document lifetime receipt of anthracycline dose
* Patient must have completed cancer treatment >= 2 years prior to study enrollment

Exclusion Criteria:

* Receiving treatment for cardiomyopathy or heart failure
* Ejection fraction of < 50% (by radionuclide angiogram or echocardiogram) or shortening fraction of < 25% (by echocardiogram)

  * Note: for instances where both are reported, and one is below the threshold, the site will have the option to re-measure it centrally at the core lab
* Uncorrected primary obstructive or severe regurgitative valvular disease:

  * Nondilated (restrictive); or
  * Hypertrophic cardiomyopathy; or
  * Significant systemic ventricular outflow obstruction
* Sustained or symptomatic ventricular dysrhythmias uncontrolled with drug therapy or implantable device
* Significant conduction defects (i.e. second or third degree atrio-ventricular block or sick sinus syndrome)
* Bradycardia: heart rate < 50 beats per minute (BPM)
* Use of an investigational drug or beta adrenergic blockers, including metoprolol, sotalol, within 30 days of enrollment
* History of drug sensitivity or allergic reaction to alpha or beta-blockers
* Low resting systolic blood pressure: < 90 mmHg
* Use of any other blood pressure lowering medication for treatment of hypertension within 30 days of enrollment except calcium channel blockers and diuretics
* History or current clinical evidence of moderate-to-severe obstructive pulmonary disease or reactive airway diseases (i.e. asthma) requiring therapy
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times upper limit of institutional normal
* Gastrointestinal, or biliary disorders that could impair absorption, metabolism, or excretion of orally administered medications
* Endocrine disorders (such as primary aldosteronism, pheochromocytoma, hyper- or hypothyroidism) not controlled with medication
* Uncontrolled diabetes (controlled diabetes per the American Diabetes Association and International Diabetes Center's Glycemic Target Goals is hemoglobin A1C < 7%)
* Anemia (hematocrit < 28%)
* Currently using select CYP2D6 inhibitor or inducer medications
* Inability to swallow pills
* Female patients who are pregnant are not eligible; women of childbearing potential require a negative pregnancy test prior to starting study drug
* Lactating females are not eligible unless they have agreed to not breastfeed their infants
* Sexually active female patients of reproductive potential are not eligible unless they agree to use an effective contraceptive method during study and for 2 months after stopping the study drug; abstinence is an acceptable method of birth control
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saro H Armenian, Principal Investigator — Children's Oncology Group
Locations (91):
- United States (86):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Mission Hospital, Asheville, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
- Australia (2):
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- IWK Health Centre, Halifax, Nova Scotia, Canada
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Armenian SH, Hudson MM, Chen MH, Colan SD, Lindenfeld L, Mills G, Siyahian A, Gelehrter S, Dang H, Hein W, Green DM, Robison LL, Wong FL, Douglas PS, Bhatia S. Rationale and design of the Children's Oncology Group (COG) study ALTE1621: a randomized, placebo-controlled trial to determine if low-dose carvedilol can prevent anthracycline-related left ventricular remodeling in childhood cancer survivors at high risk for developing heart failure. BMC Cardiovasc Disord. 2016 Oct 4;16(1):187. doi: 10.1186/s12872-016-0364-6. PMID 27716152
- See also: Pharmacologic Reversal of Ventricular Remodeling in Childhood Cancer Survivors at Risk for Congestive Heart Failure (PREVENT-CHF): A Phase IIB Randomized Placebo-Controlled Trial — https://clinicaltrials.gov/ct2/show/NCT01347970?term=NCT01347970&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 196 pts were enrolled (109 pts enrolled with Childrens Oncology Group (COG) and 87 pts enrolled on a pilot study at City of Hope (COH) 182 of those pts started tx (14 excluded: 6 ineligible and 8 pts started tx). (The (109) enrollment number in the protocol section reflects the number of pts enrolled on the COG portion of the study. Per Section 9.2 of the protocol (pt accrual and expected duration of the trial), 87 pts had already been accrued through a different mechanism the pilot study)
Groups:
- Arm I (Carvedilol): Patients receive low-dose carvedilol orally (PO) once daily (QD) or twice daily (BID) for 24 months.
Period: Overall Study
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Started | 89 | 93
2nd Timepoint Assessment of Echocardiology Required to be Analyzable (31 participants who did not have a second timepoint assessment of echocardiography were excluded, resulting in 151 analyzable participants.) | 75 | 76
Completed | 58 | 55
Not Completed | 31 | 38
Not completed — Lost to Follow-up | 5 | 8
Not completed — Pregnancy | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 20 | 20
Not completed — Relapse | 1 | 1
Not completed — Cardiac Event | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo) | Total
Number analyzed (Participants) | 89 | 93 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 74 | 77 | 151
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (10.3) | 27.7 (10.1) | 27.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 46 | 45 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 22 | 45
  Not Hispanic or Latino | 65 | 69 | 134
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 77 | 82 | 159
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 89 | 93 | 182

OUTCOME MEASURES:

1. Primary Outcome: Average Left-Ventricular Wall Thickness-Dimension Ratio Z-score (LVWT/Dz)
Description: Z-score of the ratio of left ventricular (LV) posterior wall dimension of systole to internal LV dimension in diastole, calculated for each subject by subtracting the reference healthy population mean, then dividing by the standard deviation. The Z-score indicates the number of standard deviations away from the mean of the reference population. Negative Z- score indicates worse outcome. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: We excluded 31 participants who did not have a second time point assessment of echocardiography, resulting in 151 analyzable participants.
Measure: Mean (Standard Error); unit: z-score
Groups:
- Arm I (Carvedilol): Patients received Carvedilol PO delivered at 6.25 mg twice daily (for a total dose of 12.5 mg per day) for 24 months.
- Arm II (Placebo): Patients received Placebo PO delivered at 6.25 mg twice daily (for a total dose of 12.5 mg per day) for 24 months.
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
z-score
  BL | -0.1372 (0.1711) | -0.0893 (0.1917)
  6m | -0.2167 (0.167) | 0.3215 (0.154)
  12m | -0.2416 (0.1721) | -0.2367 (0.1822)
  18m | -0.2375 (0.21) | -0.1974 (0.1976)
  24m | 0.0213 (0.2353) | -0.1834 (0.2145)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); The null hypothesis is that change in LVWT/Dz across time do not vary by arm. Assuming a type I error=0.05, 2-sided test, 15% attrition/year, and correlation range of 0.6-0.8 between measurements, we projected that a sample size of 125/arm would provide 80% power to detect an effect size of 0.23-0.32 for LVWT/Dz at 24m; Test type: Other; p = 0.15, Generalized Estimating Equation (GEE); The treatment effect was determined by testing the significance of the group by time interaction in GEE using a one degree-of-freedom (df) test; Slope = 0.163, 95% CI 2-sided [-0.057 to 0.383], Standard Error of Mean 0.112 — The treatment was considered efficacious if the group by time interaction for LVWT/Dz was statistically significant at a two-sided p<0.05 and the expected LVWT/Dz was higher for carvedilol than placebo over time

2. Secondary Outcome: Average Left Ventricular End-systolic Wall Stress
Description: Echocardiographic measure of left ventricular (LV) afterload based on LV pressure (P), volume (V), and wall thickness (T), calculated by the formula (P x V)/T, which equals the number referred to below in the Measure Type. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
g/cm^2
  BL | 93.2892 (2.222) | 90.6135 (2.9775)
  6m | 90.3088 (2.0577) | 96.8356 (2.9025)
  12m | 88.984 (2.0069) | 96.0616 (3.0406)
  18m | 93.9267 (2.4333) | 91.6458 (3.1257)
  24m | 89.2513 (2.4341) | 94.0647 (3.6562)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.03, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -3.764, 95% CI 2-sided [-7.105 to -0.424], Standard Error of Mean 1.705

3. Secondary Outcome: Average Left Ventricular End-systolic Dimension
Description: Thickness of cardiac muscle (in cm) of the left ventricle at the end of systole. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: centimeter
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
centimeter
  BL | 03.2765 (0.043) | 3.2396 (0.0459)
  6m | 3.2901 (0.0382) | 3.3023 (0.0442)
  12m | 3.262 (0.043) | 3.2964 (0.0571)
  18m | 3.32 (0.0436) | 3.2798 (0.0579)
  24m | 3.2441 (0.0435) | 3.286 (0.0607)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.05, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -0.045, 95% CI 2-sided [-0.09 to 0.001], Standard Error of Mean 0.023

4. Secondary Outcome: Average Left Ventricular End-systolic Volume
Description: The amount of blood (in ml) in the heart's left ventricle just after the heart contracts. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
ml
  BL | 42.2193 (1.3907) | 39.7354 (1.3633)
  6m | 41.6128 (1.4041) | 41.3839 (1.5337)
  12m | 42.8437 (1.3498) | 41.8113 (1.6275)
  18m | 43.1453 (1.605) | 42.5634 (2.1281)
  24m | 42.0086 (1.7268) | 42.442 (2.3661)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.17, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -2.194, 95% CI 2-sided [-5.34 to 0.951], Standard Error of Mean 1.605 — The treatment was considered efficacious if the group by time interaction for LVESV was statistically significant at a two-sided p<0.05 and the expected LVESV was lower for carvedilol than placebo over time

5. Secondary Outcome: Average Left Ventricular End-diastolic Dimension
Description: Thickness of cardiac muscle (in cm) of the left ventricle at the end of diastole. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm
Groups:
- Arm II (Placebo): Patients received Carvedilol PO delivered at 6.25 mg twice daily (for a total dose of 12.5 mg per day) for 24 months.
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
cm
  BL | 4.5836 (0.0501) | 4.5269 (0.0565)
  6m | 4.6035 (0.0431) | 4.565 (0.0463)
  12m | 4.636 (0.0556) | 4.5884 (0.0768)
  18m | 4.6032 (0.0568) | 4.5462 (0.0663)
  24 | 4.5147 (0.0614) | 4.5976 (0.067)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.01, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -0,083, 95% CI 2-sided [-0141 to -0.024], Standard Error of Mean 0.03

6. Secondary Outcome: Average Left Ventricular End-diastolic Volume
Description: The amount of blood (in ml) in the heart's left ventricle just before the heart contracts. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
ml
  BL | 99.7507 (3.0157) | 93.3155 (3.0337)
  6m | 99.3216 (2.9788) | 95.7434 (3.2631)
  12m | 102.378 (2.975) | 96.5002 (3.3889)
  18m | 101.174 (3.5977) | 99.4656 (4.0815)
  24m | 100.659 (4.0356) | 98.9602 (4.6469)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.36, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -2.397, 95% CI 2-sided [-7.499 to 2.704], Standard Error of Mean 2.603 — The treatment was considered efficacious if the group by time interaction for LVEDV was statistically significant at a two-sided p<0.05 and the expected LVEDV was lower for carvedilol than placebo over time

7. Secondary Outcome: Average Left Ventricular Mass
Description: The weight of the left ventricle adjusted for body surface area (in g/m2). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g/m^2
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
g/m^2
  BL | 57.4862 (1.2135) | 57.9322 (1.5767)
  6m | 58.2839 (1.3859) | 57.0924 (1.29)
  12m | 60.2116 (1.6786) | 59.4508 (1.4995)
  18m | 57.7053 (1.6667) | 59.1793 (1.6168)
  24m | 58.3315 (1.6478) | 59.1026 (1.8092)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.59, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 0.433, 95% CI 2-sided [-1.134 to 1.999], Standard Error of Mean 0.799

8. Secondary Outcome: Average Fractional Shortening
Description: A measure to assess preload and afterload (in %). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
percent
  BL | 28.5362 (0.4549) | 28.4339 (0.4764)
  6m | 28.5409 (0.4738) | 27.6866 (0.5799)
  12m | 29.6121 (0.483) | 28.1085 (0.4918)
  18m | 27.8219 (0.4951) | 27.8891 (0.596)
  24 | 28.0302 (0.5073) | 28.5953 (0.5901)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.84, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -0.060, 95% CI 2-sided [-0.652 to 0.532], Standard Error of Mean 0.302 — The treatment can be considered beneficial if the mean difference (treatment - control) slope is positive

9. Secondary Outcome: Average Ejection Fraction
Description: The percentage of blood leaving the heart at the end of diastole. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
Percent
  BL | 57.6 (0.69) | 57.42 (0.58)
  6m | 58.16 (0.59) | 56.84 (0.6)
  12m | 58.07 (0.62) | 56.61 (0.7)
  18m | 57.35 (0.69) | 57.6 (0.71)
  24 | 58.16 (0.79) | 57.5 (0.62)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); The null hypothesis is that change in LVEF across time do not vary by arm. Assuming a type I error=0.05, 2-sided test, 15% attrition/year, and correlation range of 1.2-1.6 between measurements, we projected that a sample size of 125/arm would provide 80% power to detect an effect size of 0.23-0.32 for LVEF at 24m; Test type: Other; p = 0.49, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 0.259, 95% CI 2-sided [-0.472 to 0.991], Standard Error of Mean 0.373 — The treatment was considered efficacious if the group by time interaction for LVEF was statistically significant at a two-sided p<0.05 and the expected LVEF was higher for carvedilol than placebo over time

10. Secondary Outcome: Average Peak Early Atrial Divided by Peak Late Atrial Velocities
Description: Ratio of peak velocity blood flow from left ventricular relaxation in early diastole (E wave) to peak velocity flow in late diastole caused by atrial contraction (A wave). "Number" shown for Unit of Measure refers to this ratio. Normal: >1. Impaired: <1. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
ratio
  BL | 1.728 (0.067) | 1.732 (0.071)
  6m | 1.642 (0.048) | 1.769 (0.069)
  12m | 1.723 (0.065) | 1.722 (0.079)
  18m | 1.732 (0.063) | 1.732 (0.081)
  24m | 1.603 (0.063) | 1.64 (0.074)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.82, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 0.009, 95% CI 2-sided [-0.065 to 0.082], Standard Error of Mean 0.038

11. Secondary Outcome: Average N-terminal Pro B-type Natriuretic Peptide
Description: B-type natriuretic peptide- a biomarker for heart failure (in pg/ml). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
pg/mL
  BL | 27.3836 (2.0697) | 31.4324 (3.424)
  6m | 31.8406 (3.3339) | 34.1857 (3.4737)
  12m | 26.8203 (3.4625) | 33.2941 (4.095)
  18m | 35.807 (3.7939) | 32.2807 (4.0405)
  24m | 34.625 (3.0875) | 33.3774 (3.6481)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.24, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 2.121, 95% CI 2-sided [-1.387 to 5.63], Standard Error of Mean 1.79 — The treatment can be considered beneficial if the mean difference (treatment - control) slope is negative

12. Secondary Outcome: Average Cardiac N-terminal Pro B-type Natriuretic Peptide
Description: N-terminal pro b-type natriuretic peptide- a biomarker for heart failure (in pg/ml). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
pg/mL
  BL | 85.6301 (13.3731) | 115.7222 (22.243)
  6m | 90.7536 (11.7877) | 128.9565 (23.736)
  12m | 87.7167 (13.38) | 115.6364 (26.823)
  18m | 99.4912 (15.7275) | 93.2105 (18.5618)
  24m | 101.8333 (14.2521) | 107.8490 (26.6515)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.55, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 5.113, 95% CI 2-sided [-11.608 to 21.835], Standard Error of Mean 8.532 — The treatment can be considered beneficial if the mean difference (treatment - control) slope is negative

13. Secondary Outcome: Average Cardiac Troponin I
Description: Troponin I is a biomarker for myocardial cell injury (in ng/ml). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
ng/mL
  BL | 0.00446 (0.0024) | 0.0011 (0.0008)
  6m | 0.00265 (0.001) | 0.00174 (0.0009)
  12m | 0.00467 (0.0014) | 0.00742 (0.0034)
  18m | 0.00737 (0.0017) | 0.00684 (0.0017)
  24m | 0.01111 (0.002) | 0.01132 (0.002)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.51, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -0.001, 95% CI 2-sided [-0.004 to 0.002], Standard Error of Mean 0.001

14. Secondary Outcome: Average Galectin-3
Description: A protein produced by activated macrophages, and a member of a family of β-galactoside-binding lectings and promotes cardiac fibroblast proliferation and collagen synthesis following myocadial injury (in ng/ml). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
ng/mL
  BL | 4.4464 (0.2625) | 5.2538 (0.6531)
  6m | 4.3252 (0.2519) | 4.3735 (0.2746)
  12m | 3.7345 (0.234) | 4.3415 (0.327)
  18m | 3.4548 (0.2482) | 4.0214 (0.2506)
  24m | 3.8073 (0.3099) | 4.0791 (0.2853)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.92, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -0.022, 95% CI 2-sided [-0.468 to 0.424], Standard Error of Mean 0.228

15. Secondary Outcome: Proportion of Patients With Reportable Adverse Events as Described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE).
Description: Patients with toxicities reported via CTEP-AERS and all Grade ≥ 2 adverse events (AEs) that can be attributed probably or definitely to the study drug are considered to have AEs. The proportion of patients with AEs are reported by arm with corresponding 95% confidence intervals.
Time Frame: From baseline to month 24 since baseline
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of patients with AE
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
Proportion of patients with AE | 0.0267 [0.0083 to 0.1125] | 0 [0 to 0.039]

16. Secondary Outcome: Average Bilirubin
Description: A liver function measurement (in mg/dL). The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
mg/dL
  BL | 0.5634 (0.0428) | 0.4989 (0.0272)
  6m | 0.5973 (0.0453) | 0.4942 (0.0262)
  12m | 0.563 (0.0487) | 0.4969 (0.0302)
  18m | 0.593 (0.0665) | 0.507 (0.04)
  24m | 0.5561 (0.0436) | 0.5449 (0.0354)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.82, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 0.024, 95% CI 2-sided [-0.18 to 0.229], Standard Error of Mean 0.104 — The treatment can be considered beneficial if the mean difference (treatment - control) slope is negative

17. Secondary Outcome: Average Aspartate Aminotransferase
Description: A liver function measurement (in U/L). Normal range is 14-20 for men, 10-36 for women. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
IU/L
  BL | 26.608 (1.726) | 25.773 (1.089)
  6m | 24.068 (1.293) | 26.342 (1.252)
  12m | 25.426 (1.423) | 27.014 (1.432)
  18m | 24.375 (1.637) | 28.411 (2.665)
  24m | 24.561 (1.488) | 27.038 (1.509)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); Test type: Other; p = 0.97, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = -0.096, 95% CI 2-sided [-4.877 to 4.685], Standard Error of Mean 2.439

18. Secondary Outcome: Average Alanine Aminotransferase
Description: A liver function measurement (in U/L). Normal range is 8-48 IU/L. The mean is reported by arm at each timepoint with corresponding standard errors.
Time Frame: Baseline before treatment, 6 months, 12 months, 18 months, 24 months after treatment initiation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
IU/L
  BL | 29.122 (2.31) | 30.467 (1.948)
  6m | 28.014 (2.533) | 32.158 (2.516)
  12m | 30.148 (2.985) | 31.155 (2.742)
  18m | 27.196 (2.645) | 30.536 (3.567)
  24m | 29.86 (3.064) | 29.245 (2.626)
Statistical Analysis 1: Comparison: Arm I (Carvedilol) vs Arm II (Placebo); The null hypothesis is that change in Average Alanine aminotransferase across time-points described above does not differ by treatment arm, tested using a longitudinal GEE analysis of Average Alanine aminotransferase with a treatment by time interaction; Test type: Other; p = 0.72, Generalized Estimating Equation (GEE); [statistical method as in outcome 1, analysis 1]; Slope = 1.248, 95% CI 2-sided [-5.595 to 8.091], Standard Error of Mean 3.491 — The treatment can be considered beneficial if the mean difference (treatment - control) slope is negative

19. Secondary Outcome: Proportion of Participants With Average Adherence > 90%
Description: The number of pills taken out of the total prescribed in a 3-month period, averaged across all study time points. The proportion of participants with average adherence rate >90% is computed by arm and corresponding 95% confidence intervals are reported.
Time Frame: Average adherence across 6 months, 12 months, 18 months, 24 months after treatment initiation are calculated.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
proportion of participants | 0.483 [0.378 to 0.588] | 0.517 [0.412 to 0.622]

20. Secondary Outcome: Proportion of Patients Who Responded "Moderately", "Quite a Bit", or "Extremely" to the Question of How Bothersome the Listed Symptom Was at Any Post-day 0 Assessment Time Point.
Description: In a questionnaire, patients responded Yes/No to certain symptoms. If answered Yes, they selected "slightly", "moderately", "quite a bit", or "extremely" regarding how bothersome the symptom was. The proportion of participants responding with any of these three categories was calculated by arm, and corresponding 95% confidence intervals are reported.
Time Frame: Responses at days 14 to 730 were combined
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
Number analyzed (Participants) | 75 | 76
Proportion of patients
  Diarrhea | 0.0533 [0.0025 to 0.1042] | 0.1316 [0.0556 to 0.2076]
  Skin rash | 0.0933 [0.0025 to 0.1042] | 0.0789 [0.0183 to 0.1396]
  Itchy skin | 0.1467 [0.0666 to 0.2267] | 0.1447 [0.0656 to 0.2238]
  Dry Mouth | 0.0667 [0.0102 to 0.1231] | 0.1711 [0.0864 to 0.2557]
  Easy bruising | 0.0133 [0 to 0.0393] | 0.0921 [0.0271 to 0.1571]
  Nosebleeds | 0.0667 [0.0102 to 0.1231] | 0.0526 [0.0024 to 0.1028]
  Sunburn easily | 0.0933 [0.0275 to 0.1592] | 0.0526 [0.0024 to 0.1028]
  Weight gain | 0.0533 [0.0025 to 0.1042] | 0.0789 [0.0183 to 0.1396]
  Fluid retention | 0.0267 [0 to 0.0631] | 0.0395 [0 to 0.0833]
  Swollen feet | 0 [0 to 0.048] | 0.0921 [0.0271 to 0.1571]
  Increased sweating | 0.0933 [0.0275 to 0.1592] | 0.0789 [0.0183 to 0.1396]
  Feeling weak in parts of your body | 0.0933 [0.0275 to 0.1592] | 0.1316 [0.0556 to 0.2076]
  Shortness of breath or wheezing | 0.0933 [0.0275 to 0.1592] | 0.0395 [0 to 0.0833]
  Chest pain or heaviness | 0.08 [0.0186 to 0.1414] | 0.0921 [0.0271 to 0.1571]
  Heart racing or skipping beats | 0.08 [0.0186 to 0.1414] | 0.0395 [0 to 0.0833]
  Feeling shaky or having tremors | 0.0533 [0.0025 to 0.1042] | 0.0789 [0.0183 to 0.1396]
  Decreased bodily movement | 0.0133 [0 to 0.0393] | 0.0395 [0 to 0.0833]
  Feeling nervous | 0.1467 [0.0666 to 0.2267] | 0.1711 [0.0864 to 0.2557]
  Feeling downhearted, sad, and/or tearful | 0.2 [0.1095 to 0.2905] | 0.1184 [0.0458 to 0.1911]
  Mood swings | 0.12 [0.0465 to 0.1935] | 0.0921 [0.0271 to 0.1571]
  Dizziness and/or lightheadedness | 0.16 [0.077 to 0.243] | 0.1316 [0.0556 to 0.2076]
  Dizziness upon standing (from sitting or lying down) | 0.1467 [0.0666 to 0.2267] | 0.1579 [0.0759 to 0.2399]
  Insomnia | 0.1733 [0.0877 to 0.259] | 0.1711 [0.0864 to 0.2557]
  Difficulty concentrating | 0.1067 [0.0368 to 0.1765] | 0.1316 [0.0556 to 0.2076]
  Interrupted sleep | 0.2 [0.1095 to 0.2905] | 0.2105 [0.1189 to 0.3022]
  Tendency to take naps | 0.12 [0.0465 to 0.1935] | 0.1053 [0.0363 to 0.1743]
  Feeling unusually tired | 0.2267 [0.1319 to 0.3214] | 0.2237 [0.13 to 0.3174]
  Falling asleep at inappropriate times | 0.0267 [0 to 0.0631] | 0.0395 [0 to 0.0833]
  Ringing in the ears | 0.0533 [0.0025 to 0.1042] | 0.0921 [0.0271 to 0.1571]
  Difficulty breathing | 0.0267 [0 to 0.0631] | 0 [0 to 0.0474]
  Sensation that I have to urinate much of the time | 0.0667 [0.0102 to 0.1231] | 0.0789 [0.0183 to 0.1396]
  Discoloration of urine (i.e., bloody) | 0 [0 to 0.048] | 0.0395 [0 to 0.0833]
  Decreased libido | 0.0667 [0.0102 to 0.1231] | 0.0526 [0.0024 to 0.1028]
  Unusually heavy menstrual flows (N/A if postmenopausal or male) | 0.2 [0.0432 to 0.3568] | 0.111 [0 to 0.230]

ADVERSE EVENTS:
Time Frame: Up to 24 months after first dose of drug
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm I (Carvedilol) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/93
Other Adverse Events (participants affected / at risk) | 2/89 | 0/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carvedilol) (N=89) | Arm II (Placebo) (N=93)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02717507/Prot_SAP_000.pdf